CLINICAL TRIAL: NCT05404542
Title: A Phase 1 Open-label Trial to Evaluate the Pharmacokinetics and Safety Following Single Dose of Tavapadon in Participants With Severe Renal Impairment Compared to Participants With Normal Renal Function
Brief Title: To Evaluate Pharmacokinetics (PK) and Safety of Tavapadon in Participants With Severe Renal Impairment Compared to Participants With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVL-751-1004
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Renal Impairment
Keywords: Healthy Volunteer; Severe Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Severe Renal Impairment (Experimental): Participants with severe renal impairment will receive a single dose of tavapadon, 0.25 milligrams (mg) tablet, on Day 1.
  Interventions: Drug: Tavapadon
- Normal Renal Function (Experimental): Participants with normal renal function will receive a single dose of tavapadon, 0.25 mg tablet, on Day 1.
  Interventions: Drug: Tavapadon

INTERVENTIONS:
Drug: Tavapadon — Oral tablets
  Other Names: CVL-751

SUMMARY:
The primary purpose is to assess the effect of renal impairment on the PK of tavapadon following administration of a single oral dose in participants with severe renal impairment relative to age, body weight, and sex-matched participants with normal renal function.

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index of ≥18.0 to 40.0 kilograms per meter square (kg/m^2), inclusive, and a total body weight >50 kilograms (kg) [(110 pounds (lbs)].
2. Age that is within ±10 years of the median age for the severe renal impairment cohort. Bodyweight that is within ±15 kg of the median bodyweight for the severe renal impairment cohort.
3. Severe renal function: estimated glomerular filtration rate (eGFR) <30 mL/min (not requiring dialysis) determined using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
4. Stable disease, defined as no clinically significant changes in disease status as documented by the most recent eGFR assessment (within at least 3 months before Screening).
5. Stable concomitant medications for the management of individual participants medical history.

Key Exclusion Criteria:

1. Serious risk of suicide in the opinion of the investigator.
2. History of substance or alcohol use disorder (excluding nicotine or caffeine) within 12 months prior to signing the informed consent form (ICF).
3. Receipt of severe acute respiratory syndrome coronavirus 2(SARS-CoV2) vaccine or booster within 7 days of planned dosing.
4. Have recently been diagnosed with symptomatic Coronavirus Disease 2019 (COVID-19) or test positive for COVID-19 within 30 days prior to signing the ICF.
5. Positive drug screen including tetrahydrocannabinol (THC).
6. Positive result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody with detectable viral ribonucleic acid (RNA) levels at Screening.
7. Positive drug screen including THC (except with a vail prescription other than medical marijuana).
8. Participants who have received an organ transplant or are currently waiting for an organ transplant and are listed on the national transplant list.
9. Participants who require dialysis.
10. Participant with nephrotic syndrome.
11. Abnormal hemoglobin.
12. Abnormal blood pressure measurement or heart rate at Screening or Check-in.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Tavapadon | pre-dose and at multiple timepoints post-dose up to Day 7
Area Under the Plasma Concentration-time Curve from Time Zero to Time t (AUC0-t) of Tavapadon | pre-dose and at multiple timepoints post-dose up to Day 7
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of Tavapadon | pre-dose and at multiple timepoints post-dose up to Day 7

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and AEs by Severity | Day 1 up to Follow-up (Day 15)
Number of Participants with Clinically Significant Abnormalities in Electrocardiogram (ECG) Values | Day 1 up to Follow-up (Day 15)
Number of Participants with Clinically Significant Abnormalities in Vital Sign Values | Day 1 up to Follow-up (Day 15)
Number of Participants with Clinically Significant Abnormalities in Laboratory Values | Day 1 up to Follow-up (Day 15)
Number of Participants with Clinically Significant Abnormalities in Physical and Neurological Examination Results | Day 1 up to Follow-up (Day 15)
Number of Participants with Change in Columbia Suicide Severity Rating Scale (C-SSRS) Score | Day 1 up to Follow-up (Day 15)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Jacksonville, Florida, Jacksonville, Florida
  - Miami, Florida, Miami, Florida
  - Tampa, Florida, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No